CLINICAL TRIAL: NCT07072845
Title: Pilot Randomized Controlled Trial to Assess the Feasibility and the Efficacy of Enhanced Brief Cognitive Behavioral Therapy (E-BCBT) for Suicidal Inpatients With Mood Disorder
Brief Title: Enhanced Brief CBT for Suicidal Inpatients With Mood Disorders
Acronym: E-BCBT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hyung Keun Park (Other)
Responsible Party: Sponsor-Investigator, Hyung Keun Park, Clinical Assistant Professor, Department of Psychiatry, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-0516
Record Dates: First submitted 2025-06-25; First posted 2025-07-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-07

CONDITIONS: Suicidal Ideation and Behaviors; Suicide Attempt; Cognitive Behavioral Therapy
Keywords: Suicidal Ideation and Behaviors; Suicide Attempt; Cognitive Behavioral Therapy for Suicidality
MeSH Terms: conditions — Suicidal Ideation; Behavior; Suicide, Attempted | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-BCBT + TAU (Experimental): Participants in this arm will receive Enhanced Brief Cognitive Behavioral Therapy (E-BCBT), a brief intervention designed for suicide prevention among psychiatric inpatients, along with treatment as usual (TAU) provided on the ward. After randomization, they will participate in five sessions of E-BCBT during hospitalization (approximately 50-60 minutes per session), in addition to receiving standard care such as pharmacotherapy, case management, and general supportive therapy offered in the inpatient setting.
  Interventions: Behavioral: Enhanced Brief Cognitive Behavioral Therapy (E-BCBT) for Suicidal Inpatients; Other: Treatment as Usual (TAU)
- TAU only (Active Comparator): Participants in this arm will receive Treatment as Usual (TAU) only. TAU is based on a short-term stabilization model and includes 24-hour multidisciplinary care delivered by an inpatient psychiatric team. Individualized treatment is provided depending on the participant's needs. TAU may include treatments such as pharmacotherapy, occupational therapy, and supportive psychotherapy, as commonly practiced in the hospital setting.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Enhanced Brief Cognitive Behavioral Therapy (E-BCBT) for Suicidal Inpatients — E-BCBT is a brief, structured cognitive behavioral therapy designed for psychiatric inpatients at risk of suicide. The primary goals are to reduce the risk of suicide attempts after discharge, improve problem-solving and coping with recent stressors related to suicidal crises, and help patients shift from maladaptive "suicidal modes" to more adaptive cognitive and behavioral patterns. The intervention consists of five individual sessions (approximately 50-60 minutes each) delivered during hospitalization. It includes two sessions on crisis management, two sessions on cognitive and behavioral strategies, and one relapse prevention session. Each session incorporates psychoeducation, skill-building, and worksheet-based self-practice to enhance self-regulation and promote continued use after discharge.
  Arms: E-BCBT + TAU
Other: Treatment as Usual (TAU) — TAU is based on a short-term inpatient stabilization model and includes 24-hour multidisciplinary care provided by the psychiatric ward. Individualized treatment may involve pharmacotherapy, occupational therapy, and supportive psychotherapy, depending on patient needs and hospital protocols.

SUMMARY:
The goal of this clinical trial is to evaluate whether enhanced brief cognitive behavioral therapy (E-BCBT) can help reduce suicidal thoughts and behaviors among psychiatric inpatients. This therapy is designed to be feasible during hospitalization and includes self-directed worksheets that may later be used independently after discharge, offering potential benefits for suicide prevention outside the hospital setting as well.

Participants will be randomly assigned to one of two groups:

* E-BCBT group: Participants will receive five sessions of cognitive behavioral therapy (approximately 50-60 minutes each) during their inpatient stay.
* TAU (treatment as usual) group: Participants will receive standard care provided on the psychiatric ward.

All participants will take part in five assessments: one before treatment, one after treatment, and three monthly follow-up assessments over the three months after discharge. Assessments include interviews, conducted in person or by phone, and questionnaires, completed online via a survey link. The entire study period will take approximately four months.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for the study:

* Hospitalized following a suicide crisis

  *A suicide crisis is defined based on the Columbia-Suicide Severity Rating Scale (C-SSRS) as meeting at least one of the following: A. A suicide attempt within 1 week prior to admission B. Current suicidal ideation and plan at the time of admission (recorded as the reason for hospitalization) and at least one prior suicide attempt within the past 2 years
* Aged 18 years or older
* Diagnosed with a depressive disorder or bipolar and related disorder based on the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) using the Mini International Neuropsychiatric Interview (M.I.N.I.) at screening
* Able to read and write in Korean without difficulty
* Capable of understanding the study procedures and providing written informed consent voluntarily

Exclusion Criteria:

Participants will be excluded if any of the following apply:

* Has an acute manic episode with psychotic features, a schizophrenia spectrum disorder, a clinically significant neurological disorder, brain injury, intellectual disability, or any other physical illness that would interfere with participation in the study.
* Receiving ongoing psychotherapy (e.g., cognitive behavioral therapy, interpersonal psychotherapy, psychodynamic psychotherapy) within 3 months prior to screening.
* Expected to be discharged within 6 working days of admission, as judged by the attending physician
* Scheduled to receive electroconvulsive therapy (ECT) during hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-04-22 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
Number of Suicide Attempts from Baseline to 3 Months After Discharge | Baseline: Within 24 hours after informed consent and within 2 days before treatment start; Post-treatment: Within 48 hours after discharge; Follow-up assessments: At 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after discharge.
  The number of suicide attempts will be assessed at five time points (baseline, post-treatment, and monthly during the 3-month follow-up) using the Columbia-Suicide Severity Rating Scale, with data cross-checked against electronic medical records.
Time to First Suicide Attempt After Discharge | 1 month, 2 months, and 3 months post-discharge
  The number of days from hospital discharge to the first reported suicide attempt, assessed through monthly follow-up interviews during the 3-month follow-up period.

SECONDARY OUTCOMES:
Intensity of suicidal ideation measured by Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline: Within 24 hours after informed consent and within 2 days before treatment start; Post-treatment: Within 48 hours after discharge; Follow-up assessments: At 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after discharge.
  Suicidal ideation intensity will be assessed using the Intensity of Ideation subscale of the C-SSRS. This clinician-administered interview includes five items (frequency, duration, controllability, deterrents, and reasons for ideation), each scored from 0 to 5. Higher scores indicate greater ideation intensity.
Severity of suicidal ideation measured by Beck Scale for Suicide Ideation (SSI) | Baseline: Within 24 hours after informed consent and within 2 days before treatment start; Post-treatment: Within 48 hours after discharge; Follow-up assessments: At 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after discharge.
  Suicidal ideation severity will be assessed using the Beck Scale for Suicide Ideation, a 19-item self-report questionnaire. Each item is scored from 0 to 2, producing a total score from 0 to 38. Higher scores indicate greater severity of suicidal ideation.
Change in depressive symptoms measured by Hamilton Depression Rating Scale (HAM-D-17) | Baseline: Within 24 hours after informed consent and within 2 days before treatment start; Post-treatment: Within 48 hours after discharge; Follow-up assessments: At 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after discharge.
  Depressive symptom severity will be assessed at five time points using the 17-item Hamilton Depression Rating Scale. This clinician-administered semi-structured interview yields total scores ranging from 0 to 52, with higher scores indicating more severe depression.
Change in depressive symptoms measured by Beck Depression Inventory-II (BDI-II) | Baseline: Within 24 hours after informed consent and within 2 days before treatment start; Post-treatment: Within 48 hours after discharge; Follow-up assessments: At 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after discharge.
  Depressive symptom severity will be assessed at five time points using the Beck Depression Inventory-II, a 21-item self-report questionnaire. Each item is scored from 0 to 3, yielding total scores from 0 to 63. Higher scores indicate greater symptom severity.
Change in hopelessness measured by the Beck Hopelessness Scale (BHS) | Baseline: Within 24 hours after informed consent and within 2 days before treatment start; Post-treatment: Within 48 hours after discharge; Follow-up assessments: At 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after discharge.
  Change in the level of hopelessness will be assessed at five time points: baseline, post-treatment, and monthly for 3 months following discharge. Hopelessness will be measured using the Beck Hopelessness Scale (BHS), a 20-item self-report questionnaire designed to assess negative expectations about the future. Each item is scored dichotomously (True/False), with total scores ranging from 0 to 20. Higher scores indicate greater levels of hopelessness and have been associated with increased suicide risk.

OTHER OUTCOMES:
Consent rate (as an indicator of feasibility) | For each participant, from the time they are found eligible through screening until the time they provide informed consent and are randomized, during the study's active recruitment period (approximately 6 months).
  Consent rate will be used as a key feasibility indicator. It is defined as the percentage of eligible participants who provided informed consent and were randomized. The rate will be calculated by dividing the number of participants who consented and were randomized by the total number of eligible participants screened during the recruitment period.
Retention rate (as an indicator of feasibility) | From randomization to each scheduled assessment point: post-treatment (within 48 hours after discharge), and 1-month (±7 days), 2-month (±7 days), and 3-month (±7 days) follow-ups after discharge, for each participant.
  Retention rate will be used as a key feasibility indicator. It is defined as the percentage of randomized participants who remained in the study and provided valid primary outcome data at each designated follow-up time point. The rate will be calculated by dividing the number of participants who completed the primary outcome assessment at each time point by the total number of participants randomized.
Adherence to treatment (as an indicator of feasibility) | From the first to the fifth scheduled treatment session, over the intervention period (approximately 7 days), for each participant assigned to the intervention group.
  Adherence to treatment will be used as a feasibility indicator. It is defined as the percentage of participants who attended all 5 scheduled treatment sessions. The rate will be calculated by dividing the number of participants who completed all sessions by the total number of participants assigned to the intervention group.
Death-Implicit Association Test (D-IAT) | Baseline: Within 24 hours after informed consent and within 2 days before treatment start; Post-treatment: Within 48 hours after discharge; Follow-up assessments: At 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after discharge.
  Implicit identification with death will be assessed using the Death-Implicit Association Test (D-IAT), a computerized task measuring automatic associations between death-related concepts and the self. The Korean version of the D-IAT, validated for local use, consists of seven blocks administered via PsychoPy software. The outcome score (D-score) is computed using a standard scoring algorithm: a positive D-score indicates a stronger implicit association between death and self, while a negative score indicates a stronger association between life and self. Higher D-scores have been associated with increased risk of suicide attempts.
Anxiety symptoms measured by the Beck Anxiety Inventory (BAI) | Baseline: Within 24 hours after informed consent and within 2 days before treatment start; Post-treatment: Within 48 hours after discharge; Follow-up assessments: At 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after discharge.
  Anxiety symptoms will be assessed at all scheduled time points using the Beck Anxiety Inventory (BAI), a 21-item self-report questionnaire. Each item is rated on a 0 to 3 scale, yielding a total score from 0 to 63. Higher scores indicate greater anxiety severity.
Emotion dysregulation measured by the Difficulties in Emotion Regulation Scale (DERS) | Baseline: Within 24 hours after informed consent and within 2 days before treatment start; Post-treatment: Within 48 hours after discharge; Follow-up assessments: At 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after discharge.
  Emotion dysregulation will be assessed at all scheduled time points using the 35-item Korean version of the Difficulties in Emotion Regulation Scale (DERS). This self-report questionnaire measures six dimensions of emotion regulation difficulties: Nonacceptance of emotional responses, Difficulties engaging in goal-directed behavior, Impulse control difficulties, Lack of emotional awareness, Limited access to emotion regulation strategies, and Lack of emotional clarity. Each item is rated on a 5-point Likert scale from 1 to 5, with higher scores indicating greater difficulties in emotion regulation.
Distress tolerance measured by the Distress Intolerance Index (DII) | Baseline: Within 24 hours after informed consent and within 2 days before treatment start; Post-treatment: Within 48 hours after discharge; Follow-up assessments: At 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after discharge.
  Distress tolerance will be assessed at all scheduled time points using the Distress Intolerance Index (DII), a 10-item self-report questionnaire. Each item is rated on a 5-point Likert scale from 0 (not at all like me) to 4 (very much like me), with total scores ranging from 0 to 40. Higher scores indicate lower distress tolerance.
Negative automatic thoughts measured by the Automatic Thoughts Questionnaire-Negative (ATQ-N) | Baseline: Within 24 hours after informed consent and within 2 days before treatment start; Post-treatment: Within 48 hours after discharge; Follow-up assessments: At 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after discharge.
  Negative automatic thoughts will be assessed using the Automatic Thoughts Questionnaire-Negative (ATQ-N), a 30-item self-report measure. Participants rate how frequently they experienced each thought on a 5-point Likert scale from 1 (not at all) to 5 (all the time). Total scores range from 30 to 150, with higher scores indicating greater frequency of negative automatic thoughts.
Positive automatic thoughts measured by the Automatic Thoughts Questionnaire-Positive (ATQ-P) | Baseline: Within 24 hours after informed consent and within 2 days before treatment start; Post-treatment: Within 48 hours after discharge; Follow-up assessments: At 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after discharge.
  Positive automatic thoughts will be assessed using the Automatic Thoughts Questionnaire-Positive (ATQ-P), a 30-item self-report measure. Each item is rated on a 5-point Likert scale from 1 (not at all) to 5 (all the time). Total scores range from 30 to 150, with higher scores indicating more frequent positive automatic thoughts.
Interpersonal needs measured by the Interpersonal Needs Questionnaire (INQ) | Baseline: Within 24 hours after informed consent and within 2 days before treatment start; Post-treatment: Within 48 hours after discharge; Follow-up assessments: At 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after discharge.
  Interpersonal needs will be assessed using the Interpersonal Needs Questionnaire (INQ), a 15-item self-report measure designed to assess two constructs: perceived burdensomeness and thwarted belongingness. Each item is rated on a 7-point Likert scale from 1 (not at all true for me) to 7 (very true for me). Higher scores reflect greater interpersonal distress.
Fearlessness about death measured by the Acquired Capability for Suicide Scale - Fearlessness About Death (ACSS-FAD) | Baseline: Within 24 hours after informed consent and within 2 days before treatment start; Post-treatment: Within 48 hours after discharge; Follow-up assessments: At 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after discharge.
  Fearlessness about death will be assessed using the Acquired Capability for Suicide Scale - Fearlessness About Death (ACSS-FAD), a 7-item self-report questionnaire. Each item is rated on a 5-point Likert scale from 0 (not at all like me) to 4 (very much like me), with higher scores indicating greater fearlessness about death.
Treatment satisfaction measured by the Client Satisfaction Questionnaire (CSQ-8) | At post-treatment (within 48 hours after discharge), for each participant in the intervention group
  Treatment satisfaction will be assessed using the Client Satisfaction Questionnaire (CSQ-8), an 8-item self-report instrument rated on a 4-point Likert scale. The measure assesses satisfaction with treatment quality, perceived effectiveness, and willingness to reuse or recommend the intervention. Higher total scores indicate greater satisfaction.
Use and perceived helpfulness of intervention techniques measured by the Utility of Techniques (UT) questionnaire | At 1-month (±7 days), 2-month (±7 days), and 3-month (±7 days) follow-up assessments after discharge, for each participant in the intervention group.
  The Utility of Techniques (UT) questionnaire will be used to assess participants' frequency of use and perceived helpfulness of specific intervention components. For each technique the participant reports having learned during the inpatient stay, they will rate frequency of use (from "not at all" to "more than 10 times per week") and helpfulness (if used, from "not at all" to "extremely"). Techniques include, for example, personalized safety planning tools and coping strategies taught during the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No